CLINICAL TRIAL: NCT06184685
Title: A Comparative Double-Blinded Randomized Study: Clinical Safety and Efficacy of Sahasthara Microemulsion Versus Diclofenac Microemulsion for Treating Primary Knee Osteoarthritis
Brief Title: Safety and Efficacy of Sahasthara ME vs Diclofenac ME for Treating Primary Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Ninnart Intharit, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ninnart Intharit 01
Record Dates: First submitted 2023-12-05; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Primary Knee Osteoarthritis
Keywords: Clinical; Topical; Microemulsion; Sahasthara; Diclofenac; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sahasthara Microemulsion (Experimental): The extract of Sahasthara remedy was obtained by maceration with 95% ethanol for 3 days. The marc was re-extracted using the same process two more times. After that, the extract was filtered, concentrated using a rotary evaporator at 40 degree C and vacuum (Rotavapor R-205, Buchi, Switzerland), to gave a yield of 10.3% w/w. Finally, SHT ethanolic extract was formulated into a microemulsion with 1% (w/w) of extract and was stored in 50 ml bottles.
  Interventions: Drug: Sahasthara Microemulsion
- Diclofenac Microemulsion (Experimental): DF-ME, which consists of 2% diclofenac sodium, was compounded according to the published instructions by RS Therapeutics Inc. (Canada) and stored in the same containers as SHT-ME.
  Interventions: Drug: Diclofenac Microemulsion

INTERVENTIONS:
Drug: Sahasthara Microemulsion — All patients were instructed to treat the knee with 2 ml, 3x/day, for 28 days. Each of the patients received the same appearance of drug packaging, which was not revealed until data analysis was completed, or medical emergency conditions would require an unblinding.
  Other Names: Diclofenac Microemulsion
  Arms: Sahasthara Microemulsion
Drug: Diclofenac Microemulsion — All patients were instructed to treat the knee with 2 ml, 3x/day, for 28 days. Each of the patients received the same appearance of drug packaging, which was not revealed until data analysis was completed, or medical emergency conditions would require an unblinding.
  Arms: Diclofenac Microemulsion

SUMMARY:
Background: Sahasthara is a traditional Thai herbal remedy used for the anti-inflammatory treatment of the musculoskeletal system, while diclofenac sodium is one of the most topically administered anti-inflammatory drug. However, there has not been scientifically researched regarding the efficacy and safety of SHT formulated as ME.

Purpose: To assess the safety and effectiveness of Sahasthara microemulsion (SHT-ME) in comparison to a diclofenac microemulsion (DF-ME) in treating primary osteoarthritis (OA) of the knee.

Methods: A randomized, double blinded clinical trial phase II was conducted. One treatment group received 1% SHT-ME, while the other received 2% DF-ME (2 ml, 3 times per day for 28 days) on their affected knee area. All patients were followed up at 14 and 28 days. Changes in the visual analogue scale (VAS) for pain as well as 100-meter walking times, the WOMAC index scores, and a global assessment were examined for efficacy. Clinical examinations, abnormalities in laboratory tests, and the incidence of adverse events (AEs) were assessed for safety.

DETAILED DESCRIPTION:
Outpatient participants, aged between 40 - 70 years old, were recruited. They were screened for symptoms of primary knee OA at the Department of Orthopedics, Thammasat University Hospital, Pathum Thani, Thailand, between October - December 2021. A diagnosis of knee OA in this clinical trial were made with a combination of clinical and radiographic findings according to the American College of Rheumatology (ACR). Inclusion criteria for participants were those who had a pain score higher than 30 mm out of 100 mm on the visual analog scale (VAS), experiencing moderate to severe pain intensity from OA in one or both knees (patients who affected by knee OA bilaterally were evaluated, which more severely affected knee was included in the study) and had OA grade 1 to 3 (moderate/medium degree of pain) according to the Kellgren-Lawrence classification grading scale for OA severity. The subjects would be excluded if they: 1) had a history of hypersensitivity to ingredients in SHT ME or DF-ME, 2) were pregnant or breast feeding, 3) had previous surgery knee replacement or intra-articular steroid injections within 3 months of inclusion in the study, 4) were having any coexisting musculoskeletal diseases (including rheumatoid arthritis, septic arthritis, metabolic arthritis, gout, pseudogout, and traumatic arthritis ) or dermatologic disorder which affected the surrounding skin of the knees, or 5) was assessed by body mass index (BMI) more than 32 kg/m2. The participants who were accepted to enroll in the study signed an informed consent.

Following enrollment, eligible patients were given a washout period of one week with no administration of analgesics before being randomly assigned to receive one of the treatments daily for 4 weeks. A randomized code number from a non-stratified randomization list generated by computer was used. The physicians, researchers, and statisticians were blinded from the allocation of patients involved in the trial. During the study, they were instructed not to use other analgesics, including injection drugs or other medications. Following the baseline visit, patients returned to the study site after 2 and 4 weeks for follow-up assessments of safety, efficacy and study protocol compliance.

In the trial, demographic data, clinical signs and symptoms, physical examination, visual analogue scale (VAS) for pain, 100-meter walk times, the WOMAC index scores (pain, physical function, stiffness), and laboratory tests (fasting blood sugar, lipid profile, liver function tests (AST, ALT, ALP), and renal function tests (BUN, creatinine clearance)) were collected as baseline data and as study data on day 14 and on day 28

ELIGIBILITY:
Inclusion Criteria:

* who had a pain score higher than 30 mm out of 100 mm on the visual analog scale (VAS)
* experiencing moderate to severe pain intensity from OA in one or both knees (patients who affected by knee OA bilaterally were evaluated, which more severely affected knee was included in the study) and had OA grade 1 to 3 (moderate/medium degree of pain) according to the Kellgren-Lawrence classification grading scale for OA severity

Exclusion Criteria:

* had a history of hypersensitivity to ingredients in SHT ME or DF-ME
* were pregnant or breast feeding
* had previous surgery knee replacement or intra-articular steroid injections within 3 months of inclusion in the study
* were having any coexisting musculoskeletal diseases (including rheumatoid arthritis, septic arthritis, metabolic arthritis, gout, pseudogout, and traumatic arthritis ) or dermatologic disorder which affected the surrounding skin of the knees
* was assessed by body mass index (BMI) more than 32 kg/m2

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
The WOMAC index | 28 days (ฺDay0, Day14, Day28)
  It is a self-administered questionnaire from the latest version of WOMAC 3.1 (the Western Ontario and McMaster Universities Osteoarthritis Index) (Haq & Davatchi, 2011; Roos et al., 1999). The patients were evaluated by the WOMAC index in terms of three domains: pain score ranged from 0 (no pain) to 4 (extreme pain); physical function score ranged from 0 (no difficulty) to 4 (the most severe difficulty); stiffness score ranged from 0 (no stiffness) to 4 (the worst stiffness).

SECONDARY OUTCOMES:
The visual analogue scale (VAS) | 28 days (ฺDay0, Day14, Day28)
  The pain intensity was measured using the visual analogue scale (VAS), a 100-mm line representing the continuum of pain degree, arranged into 3 levels of pain: mild = 0-30; moderate = 31-60; and maximum pain = 61-100 (Haefeli & Elfering, 2006).

OTHER OUTCOMES:
100-meter time walk | 28 days (ฺDay0, Day14, Day28)
  Time to walk a straight horizontal indoor distance of 100 m (100-meter time walk) and the need of the participants for taking analgesics were evaluated.
The global assessment | 28 days (ฺDay0, Day14, Day28)
  The global assessment on a 0-4 Likert scale (0: none, 4: excellent) was executed by the patients themselves at the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University, Klong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No
During publication